CLINICAL TRIAL: NCT02718716
Title: A Multicenter, Open-label, Multiple-dose Study to Evaluate the Safety, Tolerability, and Efficacy of UCB7665 in Subjects With Primary Immune Thrombocytopenia
Brief Title: Study to Evaluate Safety, Tolerability and Efficacy of UCB7665 in Subjects With Primary Immune Thrombocytopenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TP0001
Record Dates: First submitted 2016-03-11; First posted 2016-03-24 (Estimated); Results first posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2023-05

CONDITIONS: Thrombocytopenia
Keywords: ITP
MeSH Terms: conditions — Thrombocytopenia | interventions — rozanolixizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- UCB7665 4 mg/kg (Experimental): Participants in this arm received 5 subcutaneous (sc) doses of UCB7665 (rozanolixizumab) 4 milligram per kilograms (mg/kg) at 1-week intervals.
  Interventions: Drug: UCB7665
- UCB7665 7 mg/kg (Experimental): Participants in this arm received 3 sc doses of UCB7665 (rozanolixizumab) 7 mg/kg at 1-week intervals.
  Interventions: Drug: UCB7665
- UCB7665 10 mg/kg (Experimental): Participants in this arm received 2 sc doses of UCB7665 (rozanolixizumab) 10 mg/kg at 1-week intervals.
  Interventions: Drug: UCB7665
- UCB7665 15 mg/kg (Experimental): Participants in this arm received 1 sc dose of UCB7665 (rozanolixizumab) 15 mg/kg.
  Interventions: Drug: UCB7665
- UCB7665 20 mg/kg (Experimental): Participants in this arm received 1 sc dose of UCB7665 (rozanolixizumab) 20 mg/kg.
  Interventions: Drug: UCB7665

INTERVENTIONS:
Drug: UCB7665 — * Intervention Type: Biological/Vaccine
  * Pharmaceutical Form: Powder for solution for infusion
  * Concentration: 100 mg/ml - Route of Administration:
  Subcutaneous infusion
  Other Names: rozanolixizumab

SUMMARY:
The primary objective of the study is to check if an subcutaneous (sc) infusion of UCB7665 is safe and tolerated in subjects with primary immune thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of primary immune thrombocytopenia (ITP) for a minimum of 3 months prior to Screening Visit
* Subject has a platelet count <30x10^9/L at Screening and <35x10^9/L at Baseline (Visit 2)
* Subject has a current or history of a peripheral blood smear consistent with ITP
* Subject has responded to previous ITP therapy (according to the judgment of the investigator)

Exclusion Criteria:

* Subject has an immunoglobulin G (IgG) level <=6g/L at Screening Visit
* Subject has a partial thromboplastin time (PTT) >=1.5x upper limit of normal (ULN) or International Normalized Ratio (INR) >=1.5 at Screening Visit
* Subject has renal and/or liver impairment defined as:

  * Serum creatinine level of >=1.4 mg/dL for females and >=1.5 mg/dL for males at Screening Visit
* Subject has planned an elective surgical procedure in the coming 6 months
* Subject has evidence of a secondary cause of primary immune thrombocytopenia purpura
* Subject has a history of clinically relevant ongoing chronic infections
* Subject has a family history of primary immunodeficiency
* Subject has a clinically relevant active infection or has had a serious infection within 6 weeks prior to the first dose of IMP
* Subject has a history of known inflammatory bowel disease, diverticular disease, and gastric or esophageal ulceration
* Subject has experienced gastrointestinal bleed in the last 6 months prior to Screening Visit and/or has current gastritis or esophagitis
* Subject has a medical history of thrombosis
* Subject has a history of coagulopathy disorders other than ITP
* Subject has received a live vaccination within 8 weeks prior to the Baseline Visit; or intends to have a live vaccination during the course of the study or within 7 weeks following the final dose of IMP
* Subject has had prior treatment with rituximab in the 6 months prior to the Baseline Visit
* Subject has not completed the washout period for the immunosuppressants, biologics and other therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (29):
- Tp0001 1101, Adelaide, Australia
- Bulgaria (2):
  - Tp0001 1302, Pleven
  - Tp0001 1301, Sofia
- Czechia (2):
  - Tp0001 203, Olomouc
  - Tp0001 201, Prague
- Tp0001 1201, Tbilisi, Georgia
- Germany (3):
  - Tp0001 401, Berlin
  - Tp0001 403, Düsseldorf
  - Tp0001 404, München
- Italy (4):
  - Tp0001 502, Florence
  - Tp0001 506, Torino
  - Tp0001 503, Udine
  - Tp0001 505, Vicenza
- Tp0001 601, Chisinau, Moldova
- Poland (5):
  - Tp0001 702, Bialystok
  - Tp0001 703, Gdansk
  - Tp0001 701, Lodz
  - Tp0001 704, Poznan
  - Tp0001 705, Warsaw
- Romania (3):
  - Tp0001 802, Brasov
  - Tp0001 801, Bucharest
  - Tp0001 803, Craiova
- Spain (3):
  - Tp0001 902, Madrid
  - Tp0001 903, Madrid
  - Tp0001 901, Valencia
- United Kingdom (4):
  - Tp0001 1001, London
  - Tp0001 1002, London
  - Tp0001 1003, London
  - Tp0001 1004, Truro

REFERENCES:
- [Result] Robak T, Kazmierczak M, Jarque I, Musteata V, Trelinski J, Cooper N, Kiessling P, Massow U, Woltering F, Snipes R, Ke J, Langdon G, Bussel JB, Jolles S. Phase 2 multiple-dose study of an FcRn inhibitor, rozanolixizumab, in patients with primary immune thrombocytopenia. Blood Adv. 2020 Sep 8;4(17):4136-4146. doi: 10.1182/bloodadvances.2020002003. PMID 32886753
- [Derived] Smith B, Kiessling A, Lledo-Garcia R, Dixon KL, Christodoulou L, Catley MC, Atherfold P, D'Hooghe LE, Finney H, Greenslade K, Hailu H, Kevorkian L, Lightwood D, Meier C, Munro R, Qureshi O, Sarkar K, Shaw SP, Tewari R, Turner A, Tyson K, West S, Shaw S, Brennan FR. Generation and characterization of a high affinity anti-human FcRn antibody, rozanolixizumab, and the effects of different molecular formats on the reduction of plasma IgG concentration. MAbs. 2018 Oct;10(7):1111-1130. doi: 10.1080/19420862.2018.1505464. Epub 2018 Sep 12. PMID 30130439
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in March 2016 and concluded in February 2019.
Pre-assignment Details: The study included a Screening Period (1 to 28 days), a Dosing Period of 1 to 4 weeks, and an Observation Period of 8 weeks. Participant Flow refers to the Safety Set.
Period: Overall Study
Arm/Group | UCB7665 4 mg/kg | UCB7665 7 mg/kg | UCB7665 10 mg/kg | UCB7665 15 mg/kg | UCB7665 20 mg/kg
Started | 15 | 15 | 12 | 12 | 12
Completed | 14 | 15 | 12 | 12 | 12
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set which consisted of all study participants who had received at least 1 infusion (full or partial infusion) of rozanolixizumab and was used for the analysis of safety data.
Groups:
- UCB7665 4 mg/kg: Participants in this arm received 5 sc doses of UCB7665 (rozanolixizumab) 4 mg/kg at 1-week intervals.
Arm/Group | UCB7665 4 mg/kg | UCB7665 7 mg/kg | UCB7665 10 mg/kg | UCB7665 15 mg/kg | UCB7665 20 mg/kg | Total Title
Number analyzed (Participants) | 15 | 15 | 12 | 12 | 12 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 14 | 10 | 11 | 7 | 49
  >=65 years | 8 | 1 | 2 | 1 | 5 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (18.4) | 46.0 (15.9) | 46.3 (16.8) | 45.8 (14.6) | 56.1 (18.2) | 50.8 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 7 | 7 | 9 | 42
  Male | 7 | 4 | 5 | 5 | 3 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 0 | 0 | 0 | 0 | 2
  White | 13 | 15 | 12 | 12 | 12 | 64

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing at Least One Treatment Emergent Adverse Event (TEAE) During the Study
Description: TEAEs were defined as Adverse Events starting after the time of first Investigational Medicinal Product (IMP) administration up to and including 8 weeks after the final dose.
Time Frame: From Visit 2 (Week 1) until End of Study Visit or Early Termination (up to 12 weeks after the first investigational medicinal product (IMP) administration)
Population: The Safety Set (SS) consisted of all study participants who had received at least 1 infusion (full or partial infusion) of rozanolixizumab and was used for the analysis of safety data.
Measure: Number; unit: percentage of participants
Groups:
- UCB7665 4 mg/kg (SS): Participants in this arm received 5 sc doses of UCB7665 (rozanolixizumab) 4 mg/kg at 1-week intervals. Participants formed the Safety Set (SS).
- UCB7665 7 mg/kg (SS): Participants in this arm received 3 sc doses of UCB7665 (rozanolixizumab) 7 mg/kg at 1-week intervals. Participants formed the SS.
- UCB7665 10 mg/kg (SS): Participants in this arm received 2 sc doses of UCB7665 (rozanolixizumab) 10 mg/kg at 1-week intervals. Participants formed the SS.
- UCB7665 15 mg/kg (SS): Participants in this arm received 1 sc dose of UCB7665 (rozanolixizumab) 15 mg/kg. Participants formed the SS.
- UCB7665 20 mg/kg (SS): Participants in this arm received 1 sc dose of UCB7665 (rozanolixizumab) 20 mg/kg. Participants formed the SS.
Arm/Group | UCB7665 4 mg/kg (SS) | UCB7665 7 mg/kg (SS) | UCB7665 10 mg/kg (SS) | UCB7665 15 mg/kg (SS) | UCB7665 20 mg/kg (SS)
Number analyzed (Participants) | 15 | 15 | 12 | 12 | 12
percentage of participants | 80.0 | 60.0 | 58.3 | 91.7 | 100

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Week 1 until the End-of-Study Visit (8 weeks following the final dose) (up to 12 weeks after the first dose of IMP)
Arm/Group | UCB7665 4 mg/kg (SS) | UCB7665 7 mg/kg (SS) | UCB7665 10 mg/kg (SS) | UCB7665 15 mg/kg (SS) | UCB7665 20 mg/kg (SS)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/15 | 1/12 | 2/12 | 0/12
Other Adverse Events (participants affected / at risk) | 11/15 | 9/15 | 7/12 | 10/12 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UCB7665 4 mg/kg (SS) (N=15) | UCB7665 7 mg/kg (SS) (N=15) | UCB7665 10 mg/kg (SS) (N=12) | UCB7665 15 mg/kg (SS) (N=12) | UCB7665 20 mg/kg (SS) (N=12)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UCB7665 4 mg/kg (SS) (N=15) | UCB7665 7 mg/kg (SS) (N=15) | UCB7665 10 mg/kg (SS) (N=12) | UCB7665 15 mg/kg (SS) (N=12) | UCB7665 20 mg/kg (SS) (N=12)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina bullosa haemorrhagica (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (6) | 6 (7) | 3 (4) | 5 (6) | 9 (9)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT02718716/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT02718716/SAP_001.pdf